CLINICAL TRIAL: NCT03295864
Title: Arnold Chiari Malformation: the Otological Assessment as an Objective Criteria for Surgical Treatment
Acronym: MCoto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2016/36
Record Dates: First submitted 2017-09-14; First posted 2017-09-28 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Arnold-Chiari Malformation, Type 1
Keywords: Arnold-Chiari Malformation, Type 1; Multifrequency tympanometry; Inner ear pressure
MeSH Terms: conditions — Arnold-Chiari Malformation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Chiari type 1 malformation (Experimental): Tympanometry measurement at inclusion and 6 months after surgery
  Interventions: Diagnostic Test: Multifrequency tympanometry at Inclusion; Diagnostic Test: Multifrequency tympanometry 6 month after surgery
- Healthy volunteers (Experimental): Tympanometry measurement at inclusion. Every healthy volunteer will be match with a patient for his age and his BMI (body mass index).
  Interventions: Diagnostic Test: Multifrequency tympanometry at Inclusion

INTERVENTIONS:
Diagnostic Test: Multifrequency tympanometry at Inclusion — Multifrequency tympanometry measurement and particularly width of conductance tympanograms at 2 kHz will be performed for both group at inclusion
Diagnostic Test: Multifrequency tympanometry 6 month after surgery — Multifrequency tympanometry measurement and particularly width of conductance tympanograms at 2 kHz will be performed 6 months after surgery for Chiari type I malformation patient
  Arms: Patients with Chiari type 1 malformation

SUMMARY:
The aim of this study is to compare the value of multifrequency tympanometry between patients with surgical indication of treatment for a Chiari type I malformation and healthy volunteers.

DETAILED DESCRIPTION:
Prevalence of Chiari type I malformation in population is between 0.1% and 0.5%. Chiari type I malformation is responsive in perturbation of the cerebro spinal fluid flow at the cranio-cervical junction. Those perturbations caused headaches, and various otological symptoms (dizziness, tinnitus, vertigo, nystagmus, hypoacousis…). The surgical treatment consists in an occipital craniotomy to restore the cerebro spinal fluid flow at the cranio-cervical junction. Symptoms are due to increasing of the pressure in the cerebellar fossa. 81% of the patients with Chiari type 1 malformation suffer of sub clinical otological perturbations especially alteration of the vestibular test.

In the literature, hearing performance could be normalized after posterior fossa decompression. Furthermore, the multifrequency tympanometry measurement and particularly the width of conductance tympanograms at 2 kHz shows that variations of the cerebro spinal fluid pressure have consequences on the pressure of the perilymph.

Investigator's hypothesis is that tympanometry (conductance) could be an effective test to show the variation of the cerebro spinal fluid pressure.

ELIGIBILITY:
Inclusion criteria:

* Chiari type I malformation proved at MRI or CT-scan with an indication of cranio cervical decompression.
* Patients between 18 and 60 years old.
* Patient should benefit of the national health care system
* Agreement of the patient

Inclusion criteria for healthy volunteers:

* Between 18 and 60 years old.
* Free of otologic pathology
* Benefit of the national health care system
* Agreement of the volunteers

Exclusion criteria:

* Acute hydrocephaly
* Other type of Chiari disease (induced…)
* Medical history of neurosurgery
* Contraindication for MRI
* Cophosis
* Chronic otitis
* Medical history of ontological surgery
* Tympanic perforation
* Disturbance of tonal audiometry with air bone more than 20dB in 4 frequencies with abolition of stapedial reflex
* Pregnant women or nursing women
* Protected adults by French laws

Exclusion criteria for healthy volunteers:

* Medical history of neurosurgery
* Cophosis
* Chronic otitis
* Medical history of ontological surgery
* Tympanic perforation
* Disturbance of tonal audiometry with air bone more than 20dB in 4 frequencies with abolition of stapedial reflex
* Pregnant women or nursing women
* Medical history of Chiari malformation
* Chronic headaches or neck pain
* Protected adults by French laws

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Width of conductance tympanograms at 2 kHz measurement | Inclusion

SECONDARY OUTCOMES:
Multifrequency tympanometry | Inclusion and 6 months after surgery for patients with an indication of surgical management for a Chiari type I malformation
Resonance frequency | Inclusion and 6 months after surgery for patients with an indication of surgical management for a Chiari type I malformation
Audiometric parameters | Inclusion and 6 months after surgery for patients with an indication of surgical management for a Chiari type I malformation
Otological symptoms | Inclusion and 6 months after surgery for patients with an indication of surgical management for a Chiari type I malformation
Pain measurement with Headache Impact Test | Inclusion and 6 months after surgery for patients with an indication of surgical management for a Chiari type I malformation
Cerebro spinal fluid pressure of the cranio cervical junction | Inclusion and 6 months after surgery for patients with an indication of surgical management for a Chiari type I malformation

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BENARD, MD, Study Chair — USMR - CHU de Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France